CLINICAL TRIAL: NCT06879795
Title: Effect of Systemic Retinoic Acid Use on Periodontium-Related T Cell Differentiation
Brief Title: Retinoic Acid Therapy and Regulation of Salivary and Serum IL-1β, IL-8 and MCP-1 Levels
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, bestegül günay, Doctor of Dental Surgery, PhD Student, Medipol University
Other Study IDs: 1108
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acne Vulgaris; Gingivitis and Periodontal Diseases; Saliva Collection; Inflammation Biomarkers; Vitamin A
Keywords: chemokines; inflammation; periodontal health; retinoic acid; saliva
MeSH Terms: conditions — Acne Vulgaris; Gingivitis; Periodontal Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- retinoic acid users: A total of 24 periodontally healthy participants who were prescribed isotretinoin (Retinoic acid) (0.5-1 mg/kg/day) for six months to treat moderate to severe acne vulgaris or nodular acne, based on the Global Acne Grading System, were included in the study.

SUMMARY:
This prospective cohort study analysed the effects of systemic retinoic acid use on periodontal status, salivary flow rate (SFR), and salivary and serum levels of interleukin (IL)-1β, IL-8 and monocyte chemoattractant protein (MCP)-1.

DETAILED DESCRIPTION:
Vitamin A (isotretinoin, 13-cis-retinoic acid) and its metabolites are essential for various biological processes, including vision, development, and immune regulation. The periodontium, which consists of tissues supporting the teeth, can transition from health to disease due to multiple factors. The impact of retinoic acid (RA) on periodontal tissues has primarily been investigated in vitro; however, evidence suggests that it may reduce alveolar bone destruction and modulate cytokine expression, indicating potential anti-inflammatory properties. Nevertheless, there is a lack of studies examining the relationship between RA and periodontal health.

This study aims to evaluate the potential association between systemic RA use and the periodontal tissue response in terms of inflammatory markers (cytokines: IL-1β, IL-8; chemokines: MCP-1) and to assess dental/periodontal status at different time intervals. The study hypothesizes that RA use will enhance the periodontal tissue response independently of the existing bacterial biofilm and its quantity in the oral cavity, thereby negatively affecting the maintenance of periodontal health through alterations in the periodontium's defense mechanisms.

Saliva and serum samples from 24 participants were collected to assess inflammatory responses. The samples were obtained and stored at Istanbul Medipol University Mega Hospital, Turkey, and subsequently transferred to the University of Turku, Finland, for laboratory analyses. Serum and saliva samples were analyzed for inflammatory markers (IL-1β, IL-8, MCP-1) using multiplex immunoassay kits (Millipore; MILLIPLEX® Human Cytokine/Chemokine/Growth Factor Panel A-Immunology Multiplex Assay, #HCYTA-60K, Merck Millipore, Massachusetts, MA). Additionally, sociodemographic, dental, and periodontal data of each participant were analyzed.

This study will contribute to understanding the potential relationship between RA and periodontal status, as well as the effects of RA on the inflammatory response of periodontal tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Directed to use isotretinoin 0,5 to 1 mg/kg/day for 6 months for the treatment of moderate and severe acne vulgaris or nodular acne according to the global acne rating by dermatologist
2. Being at the age range of 18-30 years old
3. Willing to participate to the study
4. Periodontally Healthy

Exclusion Criteria:

1. Systemic diseases other than acne vulgaris or nodular acne
2. Use of antibiotics, anti-inflammatory drugs, nonsteroidal anti-inflammatory drugs, steroids, immunosuppressants, beta-blockers, calcium channel blockers, anticoagulants, or hormonal contraceptives within 6 months prior to the initiation of the study
3. Pregnancy or being lactating
4. Excessive use of alcohol
5. Smoking
6. Received nonsurgical periodontal therapy during preceding 6 months or surgical periodontal therapy during preceding 12 months
7. Have fewer than 20 natural teeth excluding third molars
8. Have orthodontic appliances.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient recruitment, data collection, and sample acquisition were conducted at Istanbul Medipol University, Faculty of Dentistry, and Istanbul Medipol University Mega Hospital, Dermatology Clinic, Turkey, between September 2023 and July 2024.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
bleeding on probing | at 4 time point: before retinoic acid treatment, during(6th week and 5th month) retinoic acid treatment and 2nd month after completion of retinoic acid therapy
  To assess the inflammatory status of the pocket base and pocket epithelium, bleeding was recorded 30 seconds after probing depth measurement. The presence of bleeding was scored as positive (+), while the absence of bleeding was recorded as negative (-).
  The percentage value of the Bleeding on Probing for each patient was calculated using the following formula:
  (Number of bleeding surfaces / Total number of tooth surfaces) × 100
IL-1beta, IL-8 and MCP-1 levels | at 4 time point: before retinoic acid treatment, during(6th week and 5th month) retinoic acid treatment and 2nd month after completion of retinoic acid therapy
  Interleukin(IL)-1beta, IL-8 and monocyte chemoattractant protein (MCP)-1 are inflammatory cytokines which show inflamatory changes.
salivary flow rate | at 4 time point: before retinoic acid treatment, during(6th week and 5th month) retinoic acid treatment and 2nd month after completion of retinoic acid therapy
  Salivary flow rate was calculated by the collected saliva volume SFR=Volume of saliva (mL) collected in 10 minutes/10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atalay N, Balci N, Toygar HU, Yardimci G, Gursoy UK. Serum, saliva, and gingival tissue human beta-defensin levels in relation to retinoic acid use. J Periodontol. 2023 May;94(5):597-605. doi: 10.1002/JPER.22-0466. Epub 2022 Dec 19. PMID 36440958